CLINICAL TRIAL: NCT01103635
Title: A Phase 1 Dose-Escalation Trial To Evaluate Safety, Tolerability And Immune Pharmacodynamics Of Combined Administration Of Tremelimumab (Blocking Anti-CTLA-4 Antibody) And CP-870,893 (Agonist Anti-CD40 Antibody) In Patients With Metastatic Melanoma
Brief Title: Tremelimumab and CP-870,893 in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 05609; NCI-2010-00507
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — selicrelumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive tremelimumab over 1 hour on day 1 and CD40 agonist monoclonal antibody CP-870,893 IV over 30 minutes on days 2, 22, 43, and 64. Treatment repeats every 12 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: CD40 agonist monoclonal antibody CP-870,893; Biological: tremelimumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: CD40 agonist monoclonal antibody CP-870,893 — Given IV
  Other Names: CP-870,893
Biological: tremelimumab — Given IV
  Other Names: anti-CTLA4 human monoclonal antibody CP-675,206; CP-675,206
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Monoclonal antibodies, such as tremelimumab and CD40 agonist monoclonal antibody CP-870,893, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry cancer-killing substances to them. Giving tremelimumab together with CD 40 agonist monoclonal antibody CP-870, 893 may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of giving tremelimumab together with CD40 agonist monoclonal antibody CP-870,893 in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety, dose-limiting toxicities and maximum tolerated doses of tremelimumab (administered intravenously every 12 weeks) and CP- 870,893 (administered intravenously every 3 weeks).

SECONDARY OBJECTIVES:

I To seek preliminary evidence of anti-tumor efficacy of the combination of tremelimumab and CP-870,893, including objective response rate at MTD.

II. To determine the immune pharmacodynamic changes associated with the administration of the combination of tremelimumab and CP-870,893.

OUTLINE: Patients receive tremelimumab IV over 1 hour on day 1 and CD40 agonist monoclonal antibody CP-870,893 IV over 30 minutes on days 2, 22, 43, and 64. Treatment repeats every 12 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion

* Patients with metastatic melanoma who have measurable disease
* ECOG PS 0 or 1
* Adequate bone marrow function
* WBC >= 3,000
* Hgb >= 9
* Plt >= 100
* Adequate hepatic function, defined by the following parameters:
* Total bilirubin WNL unless associated with hepatobiliary metastases or Gilbert syndrome, then total bilirubin =< 2 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN unless associated with hepatic metastases, then ALT and AST =< 5 x ULN
* Signed, written informed consent

Exclusion

* Previous treatment with any other compound that targets CD40 or CTLA4
* Concurrent treatment with any anticancer agent outside of this protocol
* Prior allogeneic bone marrow transplant
* History of brain metastases, even if previously treated
* History of autoimmune disorder, including type 1 diabetes mellitus, pemphigus vulgaris, systemic mastocytosis, systemic lupus erythromatosis, dermatomyositis/polymyositis, rheumatoid arthritis, systemic sclerosis, Sjorgen's syndrome, vasculitis/arteritis, Behcet's syndrome, autoimmune thyroiditis, multiple sclerosis, or uveitis
* History of chronic inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), celiac disease, or other chronic gastrointestinal conditions associated with diarrhea, or current acute colitis or enterocolitis of any etiology
* History of diverticulitis (even a single episode) or evidence at baseline, including evidence limited to CT scan only. Note diverticulosis is not an exclusion criterion per se.
* History (within the previous year) of stroke or transient ischemic attack, unstable angina, myocardial infarction, congestive heart failure
* History of deep venous thrombosis or migratory thrombophlebitis (Trousseau)
* Hereditary or acquired coagulopathies (e.g., hemophilia, von Willebrand's disease, or cancer-associated DIC)
* Prior allergic reactions attributed to other monoclonal antibodies
* Concurrent or planned concurrent treatment with systemic high dose (immunosuppressive) corticosteroids or treatment with systemic corticosteroids within 4 weeks of baseline
* Treatment on another therapeutic clinical trial within 4 weeks of enrollment in this trial
* Concurrent or planned concurrent treatment with anticoagulants such as Coumadin or heparin, except to maintain patency of in-dwelling catheters
* Ongoing or active infection; treatment with systemic antibiotics or antifungals for ongoing or recurrent infection (topical use of antibiotics or antifungals is allowed)
* Pregnancy or breast-feeding; female patients must be surgically sterile, be postmenopausal, or must agree to use effective contraception during the period of therapy and for 12 months following the last dose of either tremelimumab or CP-870,893; all female patients with reproductive potential must have a negative pregnancy test prior to enrollment
* Other uncontrolled, concurrent illness that would preclude study participation; or, psychiatric illness or social challenges that would entail unreasonable risk or preclude informed consent or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05-02 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by CTCAE v3.0 | 2 years
  Toxicities which occur during later cycles will be monitored and described separately. The MTD is defined as the dose level at which 0-1/6 patients experience DLT in the first 12 week cycle and at least 2/3 or 2/6 patients treated at the next higher dose level (unless MTD is level 4) experience DLT in the first 12 week cycle.
Response | 2 years
  Clinical response will be scored using RECIST criteria. Patients who do not complete a clinical response evaluation will be scored as unevaluable. The objective response rate is defined as the proportion of patients treated at the MTD who achieve either a complete or partial response. Unevaluable patients are included in the calculation of the objective response rate.
Immunological outcomes (analysis of antigen presenting cell activation, antigen-specific T cells, and tumor-specific T cells) | 2 years
  Analysis of antigen presenting cell (APC) activation, 2) analysis of antigen-specific T cells and 3) tumor-specific T cells, as described in Section 7.2. For T cell response analyses, overall immune response is defined as >2 fold pre-treatment/post-treatment increase in any of the key T cell parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vonderheide, MD, DPhil, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States